CLINICAL TRIAL: NCT01359514
Title: Mechanism-based Choice of Therapy for Neuropathic Pain: Can Treatments Success in Neuropathic Post-operative Pain be Coupled to Psychophysical Pain Modulation Profile?
Brief Title: Mechanism-based Choice of Therapy for Neuropathic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, d_yarnitsky, Head of Neurology Department, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PostOperativePain05CTIL
Record Dates: First submitted 2010-07-10; First posted 2011-05-24 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Pregabalin; Calcium Channel Blockers; Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duloxetine (Active Comparator)
  Interventions: Drug: Pregabalin
- Pregabalin (Active Comparator)
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Pregabalin — Initial dose of 75x2mg/d for one week, and then fixed dose of 150x2mg/d for the following 5 weeks
  Other Names: Calcium-channel blocker
  Arms: Duloxetine
Drug: Duloxetine — Initial dose of 30 mg/d will be given for one week, in order to minimize possible side effects and drop outs, and then a fixed dose of 60 mg/d will be given for additional 5 weeks
  Other Names: SSNRI
  Arms: Pregabalin

SUMMARY:
Mechanism-based choice of therapy for neuropathic pain:

Can treatments success in neuropathic post-operative pain be coupled to psychophysical pain modulation profile?

DETAILED DESCRIPTION:
Neuropathic or idiopathic pain patients will be assessed with the variety of pain tests including the conditioned pain modulation (CPM) and temporal summation (TS). Then, they will be offered on the double-blind design a several weeks treatment with either pregabalin or duloxetine. Patients will be followed-up weekly by phone for their pain relief and will be re-assessed in the lab toward the end of the treatment. The investigators suggest that patients with less-efficient CPM (deficient pain inhibition) will "earn" more pain relief from the treatment with duloxetine, while the patients with the enhanced pain summation will response better to pregabalin.

ELIGIBILITY:
Inclusion Criteria:

* patients planned for thoracotomy

Exclusion Criteria:

* age below 18 and above 75 years
* patients with psychiatric or cognitive dysfunction precluding use of psychophysics
* those who cannot communicate in Hebrew
* patients with existing thoracic or other current chronic pain

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
clinical pain | One year
  The pain relief will be achieved by treatment with duloxetine or pregabalin. We propose that the patients with deficient pain inhibition (As assessed by conditioned pain modulation lab test) will have better drug efficacy of cymbalta which restores the deficient level of serotonin and noradrenalin. In turn, pregabalin will be more effective in patients with enhance central sensitization of pain as measured by temporal summation assessment. In line, CPM and TS will be modulated by the treatment, in parallel with the analgesic effect.

CONTACTS AND LOCATIONS:
Overall Officials: David Yarnitsky, Professor, Principal Investigator — Rambam Health Care Campus; Michal Granot, PhD, Study Director — Haifa University
Locations (1):
- Rambam Medical center, Haifa, Israel